CLINICAL TRIAL: NCT06997302
Title: A Study on the Impact of Intelligent Nutrition Management on Clinical Outcomes in Chemotherapy Patients With Gastrointestinal Malignancies
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: TJMUCH-GI-ST01
Record Dates: First submitted 2025-03-03; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-03

CONDITIONS: Gastric (Stomach) Cancer; Esophageal Cancer
MeSH Terms: conditions — Stomach Neoplasms; Esophageal Neoplasms | interventions — Dietary Supplements

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group. (No Intervention): In the Control group, necessary nutritional support or dietary guidance were provided by clinical physicians following standard clinical procedures.
- Study group 1 (Experimental): In Research Group 1, nutritional status was assessed using a clinical nutrition analyzer, with interventions tailored to the system-generated "Nutritional Diagnosis Report" and recommendations.
  Interventions: Other: Nutritional Supplement
- Study group 2 (Experimental): Patients in Research Group 2 underwent evaluation by a multidisciplinary team comprising clinical physicians and dietitians, who collaboratively designed and delivered nutritional support.
  Interventions: Other: Nutritional Supplement

INTERVENTIONS:
Other: Nutritional Supplement — Dietary nutrition guidance.
  Arms: Study group 1; Study group 2

SUMMARY:
An increasing body of evidence suggests that nutritional status is a key factor in determining the quality of life of cancer patients. The sensitivity of cancer patients to anti-tumor treatments, the occurrence of side effects, and their quality of life are closely related to their nutritional status. Data show that about 50% of cancer patients experience a weight loss of more than 10% at the time of diagnosis and treatment, and once patients enter a cachexia state, the weight loss becomes difficult to reverse. Therefore, the extent to which nutritional interventions can impact clinical outcomes in these patients needs to be answered through clinical research. Currently, there are few studies using randomized controlled trials (RCTs) to explore how nutritional interventions can improve patients' quality of life, particularly in terms of prolonging survival. A recent RCT in a smaller sample population found that long-term, intensive, individualized nutritional counseling and support not only improved malnutrition in cancer patients, reduced treatment complications, and enhanced quality of life but also significantly extended survival time.

This study is a prospective, randomized controlled clinical trial aimed at investigating the effect of full-scale intelligent nutrition management in gastrointestinal malignancy patients (esophageal cancer, gastric cancer) undergoing chemotherapy. The study attempts to confirm that full-scale intelligent nutrition management can benefit these patients by maintaining or improving their nutritional status, and that the clinical effectiveness of intelligent nutrition management is comparable to that of professional nutritionists. This research will also provide clinical evidence for the intelligent and standardized nutritional treatment of cancer patients during the chemotherapy period.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years;
2. Voluntarily agree to participate and sign the informed consent form;
3. Diagnosed with gastrointestinal malignancy (esophageal cancer, gastric cancer) and planned to undergo chemotherapy;
4. Physical activity is acceptable, and capable of undergoing body composition analysis.

Exclusion Criteria:

1. Uncontrolled or severe heart, liver, lung, and kidney diseases;
2. History of stroke, epilepsy, or primary brain cancer, or patients with brain metastases from cancer;
3. Pregnant individuals;
4. Individuals allergic to milk, whey protein, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
European Nutritional Risk Screening (NRS) 2002 scores | 9 weeks
  NRS2002 scores for participants in all groups after 9-week nutritional intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China